CLINICAL TRIAL: NCT04326478
Title: Azithromycin Prophylaxis in Child Contacts of Cholera Patients: A Randomized Controlled Trial
Brief Title: Single Dose Azithromycin to Prevent Cholera in Children
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Jason B. Harris, MD, Chief, Division of Pediatric Global Health, Associate Professor of Pediatrics, Harvard Medical School, Attending, Pediatric Infectious Diseases, Microbiology, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020P000457
Record Dates: First submitted 2020-03-20; First posted 2020-03-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Cholera
Keywords: Cholera; Child Health
MeSH Terms: conditions — Cholera | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Each household will be randomized to either receive a single-dose of azithromycin or receive non-antibiotic placebo. All study visits after the drug administration, which occurs during the first visit, are equal for both groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin Group (Experimental): Enrolled children in a household randomized to the experimental group will receive a single weight-based dose of azithromycin administered by a trained study nurse within 12 hours of a member of their household testing positive for cholera. They will then complete 9 follow-up study visits in their home, during which rectal swabs and/or stool samples will be collected.
  Interventions: Drug: Azithromycin
- Non-antibiotic Placebo Group (Placebo Comparator): Enrolled children in a household randomized to the placebo arm will receive a single dose of non-antibiotic placebo during their first study visit, which will occur within 12 hours of a member of their household testing positive for cholera. Like the participants in the intervention arm, they will complete 9 follow-up study visits in their home, during which rectal swabs and/or stool samples will be collected.
  Interventions: Biological: Placebo

INTERVENTIONS:
Drug: Azithromycin — Enrolled children in the intervention arm of this study will receive a single weight-based dose of azithromycin (20 mg/kg, to a maximum dose of 1 gram) administered by a trained study nurse within 12 hours of a member of their household testing positive for cholera.
  Arms: Azithromycin Group
Biological: Placebo — Enrolled children in the placebo arm of this study will receive a single dose of non-antibiotic placebo administered by a trained study nurse within 12 hours of a member of their household testing positive for cholera.
  Arms: Non-antibiotic Placebo Group

SUMMARY:
This study aims to determine whether single-dose azithromycin is effective in preventing cholera in children who are at extremely high risk of infection. The study will also determine the effect of this intervention on the development of antibiotic resistant bacteria. The results will inform future strategies to prevent cholera in children, and improve overall understanding of the impact of azithromycin on antibiotic resistance.

DETAILED DESCRIPTION:
Vibrio cholerae causes 3 million cases of cholera and 100,000 deaths annually. An ongoing epidemic in Yemen has caused 1.7 million cases of cholera, with 58% of cholera-related deaths occurring in children. The World Health Organization (WHO) has targeted the elimination of cholera transmission by the year 2030, but the increasing burden of cholera suggests that more effective approaches are needed to prevent the disease. Access to safe water and sanitation and the use of oral cholera vaccines (OCV) are central to the WHO-proposed approach, but children remain particularly vulnerable. Children are at the highest risk of severe disease, and current cholera vaccines are ineffective in young children. In addition, natural disasters and human conflict often delay vaccination and other large-scale interventions.

Effective antibiotics reduce the volume and duration of diarrhea in cholera by over 50% and bacterial shedding by 80%. They are recommended for the treatment of moderate to severe cholera. Due to limited data, there are no standards for the use of antibiotic prophylaxis for cholera, resulting in widely varied clinical practices and the frequent use of antibiotics with unproven efficacy. For this reason, the WHO Global Task Force on Cholera Control has prioritized research in this area, suggesting that further use of prophylactic antibiotics for cholera should be stopped until prospective studies designed to measure the effectiveness of antibiotic prophylaxis and its impact on antibiotic resistance can be conducted. This study will address these two knowledge gaps. This study will determine whether a single dose of azithromycin is effective in preventing V. cholerae infection in children, and evaluate the impact of its administration on antibiotic resistance in the gut. This study focuses on children because current OCVs are ineffective in young children and because children are at the highest risk of infection and mortality from cholera. While single-dose azithromycin is a preferred treatment for cholera, it has never been studied as prophylaxis. Azithromycin has also been shown to be safe and beneficial in other recent chemoprophylaxis studies in children.

This is a double-blinded cluster randomized clinical trial of single-dose azithromycin to prevent cholera in children who are household contacts of a patient with cholera in Dhaka, Bangladesh. 920 children ages 1-15 years from 400 households in Dhaka, Bangladesh, who have shared cooking facilities for the prior three days with a household member with moderate to severe V. cholerae O1 infection, can participate in this study.

ELIGIBILITY:
Inclusion criteria:

* Shared cooking facilities for the prior three days with a household member who tested positive for cholera
* Age 1 to 15 years
* A parent or guardian available to provide informed consent
* Intention to remain enrolled in the study for 6 months

Exclusion criteria:

* Participation in any other drug, device, or vaccine trial at present or within the past 30 days
* Known or suspected hypersensitivity to azithromycin or other macrolide antibiotics

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 920 (Estimated)
Dates: Start 2021-10-31 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of V. cholerae infection in household contacts of cholera index cases | 57 months after enrollment of first subject
  The presence of V. cholerae O1 will be determined via the culturing of specimens collected via rectal swab sampling. Rectal swab acquisition will begin on the day of azithromycin administration and repeat on days 2, 3, 5, 6, and 7 following the intervention.

SECONDARY OUTCOMES:
Duration of V. cholerae shedding | 50 months after enrollment of first subject
  Duration of shedding will be assessed via quantitative polymerase chain reaction (qPCR) following rectal swab specimen collection during the first week following azithromycin administration. Duration of V. cholerae shedding (Ds) is defined as the number of days of in which a rectal swab culture is positive during the first week of follow-up.
Presence of any antibiotic or its metabolite detected by liquid chromatography-mass spectrometry (LC/MS) in the stool, beyond the assigned azithromycin intervention | 50 months after enrollment of first subject
  The impact of single-dose azithromycin use on use of other antibiotics compared to education alone will be assessed via enhanced antimicrobial resistance (AMR) metagenomics following stool collection once during the first week following azithromycin intervention as well as at the 1- and 6-month study visits.
Rate of acquisition of antibiotic resistance following azithromycin treatment | 50 months after enrollment of first subject
  The presence or absence of azithromycin immediate- or resistant-V.cholerae isolates, macrolide resistance genes in the intestinal metagenome, and clinically relevant AMR genes to the six major antibiotic classes in overall gut microbiota will be assessed via AMR-metagenomics performed on specimens collected via rectal swab collection at each study visit, and via stool collection on the fourth day following azithromycin administration as well as at the 1- and 6-month study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jason B Harris, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- icddr,b Dhaka hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No